CLINICAL TRIAL: NCT04767360
Title: Short-term Therapeutic Effects of Functional Electrical Stimulation Device Bioness L300 on the Somatosensory Cortical Representation in the Rehabilitation of Patients After Stroke
Brief Title: Effects of BIONESS in Rehabilitation of Stroke
Acronym: EFES-BIO-SEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LMU Klinikum (Other)
Collaborators: Peter Young Neurological Clinic Medicalpark Bad Feilnbach, Germany (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Benedikt Schoser, Senior consultant neurologist, LMU Klinikum
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BFB-FBI-001
Record Dates: First submitted 2021-02-17; First posted 2021-02-23 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: clinical sequential two-period crossover-design study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open labele BIONESS-Training (Other): Four-week therapeutic treatment of foot drop with the electrical stimulation device Bioness L300. This treatment will be performed five times a week for at least 30 minutes
  Interventions: Device: Bioness-300

INTERVENTIONS:
Device: Bioness-300 — Therapeutic treatment of foot drop with the electrical stimulation device Bioness L300.

SUMMARY:
A four-weeks randomized clinical two-period crossover-design study will be conducted. Each patient will be randomized in a two separate consecutive treatment periods (Parallel Group Design). "Group A" will be treated with functional electrical stimulation (FES) and a second "Gruppe B" will be treated without FES for two weeks. After this period Group A and Group B will switched.

DETAILED DESCRIPTION:
Prediction of motor recovery in the upper-limb (UL) / lower-limb (LL) in patients with stroke is generally based on clinical examination. However, according to former studies neurophysiological measures may also have a predictive value. In the acute phase, the combination of the motor score and SEPs are best predictive of outcome. Neurophysiological measures alone are of limited value in predicting long term outcome. However, predictive accuracy is substantially improved through the combined use of both of these measures and clinical variables.

A four-weeks randomized clinical two-period crossover-design study will be conducted. Each patient will be randomized in a two separate consecutive treatment periods (Parallel Group Design). "Group A" will be treated with functional electrical stimulation (FES) and a second "Gruppe B" will be treated without FES for two weeks. After this period Group A and Group B will switched.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 18 and 75
* Inadequate ankle dorsiflexion during the swing phase of gait, resulting in inadequate limb clearance
* Medically stable for at least one week following the last episode of stroke
* Stable medication for four weeks
* Adequate cognitive and communication function to give informed consent, understand the training instructions, use the device, and give adequate feedback
* Ability to walk with or without an assistive device (except parallel bars) at least 10 meters

Exclusion Criteria:

* • Lower motor neuron injury with inadequate response to stimulation

  * History of falls greater than once a week
  * Severe cardiac disease such as myocardial infarction, congestive heart failure, or a demand pacemaker
  * Patients who have other electrical stimulation devices implemented
  * Patients with epilepsy and with autoimmune diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
SEP measurement | 4 weeks
  in improving pathological latencies and / or amplitudes of somatosensory evoked potentials (SEPs)
  • N35, P40, N50 (lower limb / tibial nerve) amplitude of somatosensory evoked potential [ Time Frame: Change from baseline at 4 weeks]

SECONDARY OUTCOMES:
Motor score improvement | 4 weeks
  • Dorsal flexion/plantar extension of the ankle strength will be measured by Janda's classification of muscle imbalance patterns (Force produced by voluntary dorsiflexion). [ Time Frame: Change from baseline at 4 weeks]

CONTACTS AND LOCATIONS:
Overall Officials: Benedikt Schoser, MD, Principal Investigator — Friedrich-Baur-Institute, Dep. of Neurology LMU Klinikum Munich Germany
Locations (1):
- Neurological Clinic Medicalpark Bad Feilnbach, Bad Feilnbach, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mijic M, Schoser B, Young P. Efficacy of functional electrical stimulation in rehabilitating patients with foot drop symptoms after stroke and its correlation with somatosensory evoked potentials-a crossover randomised controlled trial. Neurol Sci. 2023 Apr;44(4):1301-1310. doi: 10.1007/s10072-022-06561-3. Epub 2022 Dec 21. PMID 36544079
- See also: homepage Medicalpark Clinics — http://www.medicalpark.de